CLINICAL TRIAL: NCT02147080
Title: A Tailored Internet Intervention to Reduce Skin Cancer Risk Behaviors Among Young Adults
Acronym: UV4me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carolyn Heckman, Associate Professor, Fox Chase Cancer Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CA154928-01 (NIH); 1R01CA154928 (NIH)
Record Dates: First submitted 2014-05-22; First posted 2014-05-26 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Skin Neoplasms
Keywords: prevention or control
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tailored Intervention (Experimental): Subject has access to the tailored web intervention
  Interventions: Behavioral: UV4me
- Skin Cancer Foundation Website (Active Comparator): Subject has access to the pre-existing Skin Cancer Foundation website
  Interventions: Behavioral: Skin Cancer Foundation website
- Assessment Only Condition (No Intervention): Subjects will only complete assessments

INTERVENTIONS:
Behavioral: UV4me — Tailored website includes: personalized responses to quizzes, information on skin type and burn risk, UV damage photo of similar individual, avatar activity, age progression images, personal risk calculator, SPF (sun protection factor) calculator
  Other Names: Tailored Intervention for Skin Cancer Risk Reduction
  Arms: Tailored Intervention
Behavioral: Skin Cancer Foundation website — Current best practice website for skin cancer and prevention. Includes information, images, news, and opportunities for advocacy.
  Arms: Skin Cancer Foundation Website

SUMMARY:
Skin cancer is the most common cancer in the US, with over a million new cases diagnosed yearly. Young adults are increasingly at risk of melanoma. Contributing to the increasing skin cancer risk is the fact that US adolescents have the lowest skin protection rates of all age groups and also demonstrate increased exposure to natural and artificial UV radiation. Innovative interventions are needed to have an impact on skin cancer risk among young people. Unlike previous interventions, our skin cancer risk reduction intervention will be tailored (or personalized) to each individual participant and delivered via the Internet. The intervention will emphasize appearance concerns, which are known to be the primary motivation for UV exposure and lack of skin protection among young adults. This will be accomplished in part through the use of personalized facial images showing UV damage as well as computerized age progression demonstrations.

Primary Aim 1. To examine the efficacy of a tailored intervention delivered via the Internet designed to increase skin protection and decrease sun exposure behavior among young adults at moderate to high risk of developing skin cancer. Participants will be randomized to the tailored intervention, the Skin Cancer Foundation website, or an assessment only condition.

Aim 2. To evaluate whether sociodemographic variables (sex, race/ethnicity, skin type, family history of skin cancer), appearance consciousness, and past exposure and protective behaviors moderate intervention effects.

Aim 3. To evaluate whether Integrative Model constructs (UV-related knowledge, risk perception, beliefs, norms, self-efficacy, and intentions) mediate intervention effects.

The goals of future research would be to enhance the tailored intervention, for example, by adding additional contacts or Internet technologies or features, disseminate the intervention, assess the longevity of effects, and/or adapt the tailored intervention for use with other cancer risk behaviors or at risk groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25 years old
* Moderate to high risk of skin cancer (cut-off of >=27 on the Brief Skin Cancer Risk Assessment Tool)

Exclusion Criteria:

* History of skin cancer

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1234 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Sun protection | Follow-up 1 (3 weeks after baseline)
  Continuous measure examining frequency of sun protection behaviors (e.g., sunscreen use, clothing, shade, sunglasses), using items adapted from Glanz and colleagues (2008)
Sun protection | Follow-up 2 (12 weeks after baseline)
  Continuous measure examining frequency of sun protection behaviors (e.g., sunscreen use, clothing, shade, sunglasses), using items adapted from Glanz and colleagues (2008)
Outdoor UV Exposure | Follow-up 1 (3 weeks after baseline)
  How many hours participants spend in the sun during peak daylight hours during the week
Outdoor UV exposure | Follow-up 2 (12 weeks after baseline)
  How many hours participants spend in the sun during peak daylight hours during the week

SECONDARY OUTCOMES:
Indoor Tanning | Follow-up 1 (3 weeks after baseline)
  Number of indoor tanning sessions in past month
Indoor Tanning | Follow-up 2 (12 weeks after baseline)
  Number of indoor tanning sessions in past month

OTHER OUTCOMES:
Spray-on tan | Follow-up 1 (3 weeks after baseline)
  Number of spray-on tanning sessions in past month
Spray-on tan | Follow-up 2 (12 weeks after baseline)
  Number of spray-on tanning sessions in past month
Sunless tanning creams | Follow-up 1 (3 weeks after baseline)
  Number of times sunless tanning cream has been used in the past month
Sunless tanning creams | Follow-up 2 (12 weeks after baseline)
  Number of times sunless tanning cream has been used in the past month

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Heckman, Ph.D, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Heckman CJ, Handorf EA, Darlow SD, Ritterband LM, Manne SL. An online skin cancer risk-reduction intervention for young adults: Mechanisms of effects. Health Psychol. 2017 Mar;36(3):215-225. doi: 10.1037/hea0000420. Epub 2016 Nov 7. PMID 27819460
- [Derived] Heckman CJ, Darlow SD, Ritterband LM, Handorf EA, Manne SL. Efficacy of an Intervention to Alter Skin Cancer Risk Behaviors in Young Adults. Am J Prev Med. 2016 Jul;51(1):1-11. doi: 10.1016/j.amepre.2015.11.008. Epub 2016 Jan 22. PMID 26810358